CLINICAL TRIAL: NCT02254356
Title: Zilver PTX Post-Market Surveillance Study of Bare Metal Stents for Treating Femoropopliteal Artery Disease in Japan
Brief Title: Zilver Flex Post-Market Study in Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-005-FLX
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Peripheral Arterial Disease (PAD)
Keywords: drug-eluting stent, paclitaxel-eluting stent, peripheral artery disease, peripheral vascular disease, superficial femoral artery, popliteal artery
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

ARMS (1):
- Zilver (Experimental)
  Interventions: Device: Zilver Flex Bare Metal Stent

INTERVENTIONS:
Device: Zilver Flex Bare Metal Stent

SUMMARY:
Japanese post market clinical study of the Zilver Flex device.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic peripheral arterial disease (PAD) involving the above-the-knee femoropopliteal arteries

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2012-05; Primary Completion 2017-12-26 (Actual); Study Completion 2017-12-26 (Actual)

PRIMARY OUTCOMES:
Occurrence of stent fracture | 3 years
Rate of adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Dake, MD, Principal Investigator — Department of Cardiothoracic Surgery, Stanford University Medical Center, Stanford, CA
Locations (1):
- Fukuoka Sanno Hospital, Fukuoka, Japan